CLINICAL TRIAL: NCT02136355
Title: A Phase II Trial Measuring the Integration of Stereotactic Radiotherapy Plus Surgery in Early Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MISSILE NSCLC
Record Dates: First submitted 2014-05-08; First posted 2014-05-13 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Body Radiation Therapy plus Surgery (Experimental): Stereotactic body radiation therapy followed by surgical resection
  Interventions: Radiation: Stereotactic Body Radiation Therapy plus Surgery

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy plus Surgery — Stereotactic body radiation therapy followed by surgical resection

SUMMARY:
Stereotactic ablative radiotherapy (SABR) is a new radiation treatment that delivers high-dose, precise radiation to small tumors in 1-3 weeks of treatment.

The study combines SABR and surgery to treat non-small cell lung cancer. SABR will be done first, with surgery done approximately 10 weeks later. There will be some extra imaging done before and after the SABR.

The purpose of this study is to determine how effective SABR is in killing the cancer cells, and if SABR can help make surgery more effective.

DETAILED DESCRIPTION:
The advent of stereotactic ablative radiotherapy (SABR) has provided a novel, promising treatment for patients with early-stage non-small cell lung cancer. SABR uses modern radiotherapy planning and targeting technologies to precisely deliver larger, ablative doses of radiotherapy.

The use of SABR as neoadjuvant therapy prior to surgery may provide a novel therapeutic opportunity. In oncology, the use of neoadjuvant radiotherapy or chemoradiotherapy prior to surgery has become widespread for several types of cancer, and in many instances improves local control over and/or survival compared to surgery alone. Neoadjuvant radiotherapy provides several theoretical advantages, including potentially decreasing the rate of positive margins, decreasing the size of the required resection, or by sterilizing the tumor to avoid seeding of circulating tumor cells during surgery. Although radiologic outcomes after SABR illustrate local control rates of approximately 90% in many studies, the presence of residual post-treatment fibrosis may confound this assessment of recurrence.

The goal of this study is to evaluate a novel treatment approach: the combination of neoadjuvant SABR followed by surgical resection in patients with T1T2N0 non-small cell lung cancer, in order to measure the true pathologic rates of local control after SABR, to develop new imaging biomarkers or response, and to assess clinical outcomes, including toxicity, relapse patterns, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* Histologically confirmed non-small cell lung cancer
* Tumor stage T1 or T2a (less than or equal to 5 cm)
* No evidence of nodal disease (N0)
* No evidence of distant metastases (M0)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 Life expectancy > 6 months
* Adequate forced expiratory volume at one second (FEV1), defined as a predicted post-operative FEV1 of 30% or greater

Exclusion Criteria:

* Serious medical comorbidities or other contraindications to radiotherapy or surgery
* Prior history of lung cancer within 5 years
* Prior thoracic radiation at any time
* Inability to attend full course of radiotherapy, surgery, or follow-up visits
* Contrast allergy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Tumor response | 2.5 years
  Percentage of patients who exhibit a lack of viable tumor after surgical resection

SECONDARY OUTCOMES:
Predictive value of imaging biomarkers | 2.5 years
  Predictive value of novel imaging biomarkers compared to pathologic outcome (complete response or non-complete response to treatment)
Tumor recurrence | 7 years
  Time to local recurrence, regional recurrence, and distant recurrence of disease will be measured
Toxicity of the combined approach of SABR + surgery | 7 years
  Toxicity of the combined approach of SABR plus surgical resection will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Quality of life measures , including physical well-being, functional well-being, and lung-cancer subscale questions | 7 years
  The FACT-TOI is a summary score derived from the FACT-L and is composed of 21 items, including physical well-being, functional well-being, and lung-cancer subscale questions

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, PhD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada

REFERENCES:
- [Derived] Yang DM, Palma DA, Kwan K, Louie AV, Malthaner R, Fortin D, Rodrigues GB, Yaremko BP, Laba J, Gaede S, Warner A, Inculet R, Lee TY. Predicting pathological complete response (pCR) after stereotactic ablative radiation therapy (SABR) of lung cancer using quantitative dynamic [18F]FDG PET and CT perfusion: a prospective exploratory clinical study. Radiat Oncol. 2021 Jan 13;16(1):11. doi: 10.1186/s13014-021-01747-z. PMID 33441162
- [Derived] Palma DA, Nguyen TK, Louie AV, Malthaner R, Fortin D, Rodrigues GB, Yaremko B, Laba J, Kwan K, Gaede S, Lee T, Ward A, Warner A, Inculet R. Measuring the Integration of Stereotactic Ablative Radiotherapy Plus Surgery for Early-Stage Non-Small Cell Lung Cancer: A Phase 2 Clinical Trial. JAMA Oncol. 2019 May 1;5(5):681-688. doi: 10.1001/jamaoncol.2018.6993. PMID 30789648
- [Derived] Palma DA, Nguyen TK, Kwan K, Gaede S, Landis M, Malthaner R, Fortin D, Louie AV, Frechette E, Rodrigues GB, Yaremko B, Yu E, Dar AR, Lee TY, Gratton A, Warner A, Ward A, Inculet R. Short report: interim safety results for a phase II trial measuring the integration of stereotactic ablative radiotherapy (SABR) plus surgery for early stage non-small cell lung cancer (MISSILE-NSCLC). Radiat Oncol. 2017 Jan 27;12(1):30. doi: 10.1186/s13014-017-0770-7. PMID 28129789